CLINICAL TRIAL: NCT04917406
Title: Randomized Clinical Trial: Comparison in the Treatment of Plantar Fasciitis by Iontophoresis Versus Ultrasound.
Brief Title: Effect of Iontophoresis vs. Ultrasound and Iontophoresis in Plantar Fasciitis". Plantar Fasciitis"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Aurora Castro-Méndez, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US-Foot 3
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Iontophoresis; Ultrasound Therapy; Complications; Fasciitis, Plantar; Pain, Acute
MeSH Terms: conditions — Fasciitis, Plantar; Acute Pain | interventions — Dexamethasone; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of iontophoresis (Experimental): Lidocaine (local anesthetic) associated with dexamethasone (corticosteroid) will be administered by iontophoresis technique. Dose per session and iontophoresis: 10 minutes with an intensity of 4 mA.
  Interventions: Drug: Application of lidocaine together with dexamethasone
- Use of ultrasound (Active Comparator): The treatment for the control group will be applied with a frequency of 3 times a week as usually performed in the ACP of the University of Seville. The application dose will be 0.65 Watt for 7 minutes in the area of most painful affectation by means of a circular movement and 1MZ head.
  Interventions: Device: Application of ultrasound as physical therapy

INTERVENTIONS:
Drug: Application of lidocaine together with dexamethasone — Lidocaine 2% is applied on the positive pole while dexamethasone 4 mg/ml is applied on the negative pole. Through the use of current the drugs penetrate the fascia.
  Arms: Use of iontophoresis
Device: Application of ultrasound as physical therapy — The application dose will be 0.65 Watt for 7 minutes in the area of most painful affectation by means of a circular movement and a 1MZ head.
  Arms: Use of ultrasound

SUMMARY:
Plantar fasciitis is inflammation of plantar fascia.The main symptom of plantar fasciitis manifests itself as localized pain in the inner area of the foot and increases in intensity after long periods of standing or resting. Its etiology is multifactorial and risk factors include overweight, female gender, physical exercise (impact sports), biomechanical imbalances of the foot and possible dysfunction of the functional twin-ankle-plantar system.Generally speaking, conservative measures are recommended as initial treatment for plantar fasciitis, and in situations where these are ineffective, corticosteroids are sometimes administered. At the local level, the route of administration can be by infiltration or iontophoresis.Iontophoresis consists of administering a drug through the skin by applying an electric current locally. This technique can be considered as a safe and effective method within the SLTF (Transcutaneous Drug Delivery Systems). It consists of introducing ions through the skin by means of electricity using a direct current, with an electrode carrying a positive charge (anode) and a negative charge (cathode). Its administration is produced thanks to the repulsive force to carry the compound through the skin by means of galvanic current.

This study aims to assess whether treatment with iontophoresis in subjects with plantar fasciitis can show a more positive evolution in pain after a 6-week treatment period (treatment frequency: 1 time per week) versus ultrasound (3 times per week) for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* plantar fasciitis
* fascia thickness (greater or equal to 4mm).

Exclusion Criteria:

* skin lesion
* sensory neuropathy
* current use of plantar supports
* taking pharmacological treatment (15 days) or previous infiltrations (6 months)
* previous surgery or fractures of the lower limb
* pregnancy
* allergy to the applied drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Fasciitis pain | Baseline
  Visual analog scale VAS to evaluate Heel pain intensity was referred to as 0-10, in which 0= no pain at all and 10= the worst pain possible
Health status | Baseline
  EQ-5D assesses health status in terms of five dimensions of health and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. EQ-5D can also be referred to as a patient-reported outcome (PRO) measure, because patients can complete the questionnaire themselves to provide information about their current health status and how this changes over time. 'EQ-5D' is not an abbreviation and is the correct term to use when referring to the instrument in general
Plantar fascia thickness in mm | Baseline
  The plantar fascia is assessed by ultrasound.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement PGI-I questionnaire | 1 month
  Patient (PGI-I). Patient Global Impression of Improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol